CLINICAL TRIAL: NCT02909738
Title: Measuring Ability of Healthy Volunteers to Power a Bicycle-powered Oxygen Concentrator
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Lara Brewer, Ph.D., University of Utah
Other Study IDs: IRB_00089531
Record Dates: First submitted 2016-09-16; First posted 2016-09-21 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Physical Exertion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Volunteers: Healthy volunteers willing to pedal a bike for 30 minutes.
  Interventions: Other: Volunteer to pedal a bicycle

INTERVENTIONS:
Other: Volunteer to pedal a bicycle

SUMMARY:
The investigators would like to test how well healthy human volunteers power a modified oxygen concentrator. The investigators modified the oxygen concentrator to be powered by a bicycle instead of wall power so that it can be used in low resource countries where the power supply is unreliable.

DETAILED DESCRIPTION:
The investigators would like to test how many healthy people can power the oxygen concentrator by pedaling the bike for at least 30 minutes. If the healthy volunteers can bike for at least 30 minutes, the investigators assume they are pedaling at or below their lactate threshold. The investigators have literature values which suggest bigger people should be able to output more work, and the investigators wish to use a sample of the population to verify that most of the people can power our system. The investigators have a good estimate of the power required by our system, and the investigators want to verify the average person can actually do what we calculated is necessary.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers will be included if they are between 18 and 45 years of age and if they do not have physical restrictions which would preclude them from riding a bike for 30 minutes.

Exclusion Criteria:

* 1)anyone with known cardiovascular, pulmonary, or metabolic disease or

  2)an age of greater than 45 or

  3) one or more of the following symptoms:
  * On medication for their heart
  * Suffer from pains in their chest
  * Ever feel faint of have spells of severe dizziness
  * High blood pressure
  * Currently on blood pressure medication
  * Have a bone or joint problem such as arthritis that has been aggravated by exercise
  * Unaccustomed to vigorous exercise
  * Have experienced unusual heart beats such as skipped beats or palpitations
  * Experience shortness or loss of breath while walking with others your own age
  * Have been diagnosed with diabetes

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-08; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Capable of pedaling the bike for 30 minutes | 30 minutes from the start time
Average heart rate | Average for the 30 minute pedaling session
volume of oxygen generated | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No